CLINICAL TRIAL: NCT04017819
Title: Biodistribution and Pharmacokinetic Study of the Positron Emission Tomography (PET) Radiopharmaceutical [18F]-C-SNAT4
Brief Title: Biodistribution&Pharmacokinetic of Position Emission Tomography(PET) Radiopharmaceutical 18F C SNAT4
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: funding
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-49038; LUN0108 (Other: OnCore); IRB-49038 (Other: Stanford IRB)
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Positron-Emission Tomography; Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Healthy volunteers (Group 1) (Active Comparator): Group 1(n = 5) healthy volunteers. Each participant in this part of the study will receive a single dose of [18F]-C-SNAT4 and then undergo three times of whole body (WB) PET/CT scans (Scan 1: 60 minutes dynamic scan; Scan 2: WB skull base-thigh at 90 minutes +/- 10 minutes post injection; Scan 3: WB skull base-thigh at 120 minutes +/- 10 minutes post-injection of [18F]-C-SNAT4).
  Interventions: Drug: 18F-C-SNAT4; Device: Positron emission tomography (PET)/Computed tomography (CT) Scan
- Patients with newly diagnosed lung cancer (Group 2) (Experimental): Group2 (n = 5) newly diagnosed lung cancer. Each participant in this part of the study will receive a single dose of [18F]-C-SNAT4 and then undergo three times of whole body (WB) PET/CT scans (Scan 1: 60 minutes dynamic scan; Scan 2: WB skull base-thigh at 90 minutes +/- 10 minutes post injection; Scan 3: WB skull base-thigh at 120 minutes +/- 10 minutes post-injection of [18F]-C-SNAT4).
  Interventions: Drug: 18F-C-SNAT4; Device: Positron emission tomography (PET)/Computed tomography (CT) Scan
- Patients with lung cancer undergoing non-surgical tx (Group 3) (Experimental): Group 3 (n = 10) lung cancer after non-surgical therapy. Each participant in this part of the study will receive a total of 2 doses of [18F]-C-SNAT4 (on 2 separate occasions spaced at least 1 week apart, each of which will be followed by undergoing a [18F]-C-SNAT4 PET/CT scan)
  Interventions: Drug: 18F-C-SNAT4; Device: Positron emission tomography (PET)/Computed tomography (CT) Scan

INTERVENTIONS:
Drug: 18F-C-SNAT4 — Radiotracer- Dose 10 mCi
Device: Positron emission tomography (PET)/Computed tomography (CT) Scan — Positron emission tomography (PET)/Computed tomography (CT) Scan

SUMMARY:
Primary Objectives

* Determine the biodistribution of [18F]-C-SNAT4 in 5 healthy volunteers. Secondary Objectives
* Determine the dosimetry of [18F]-C-SNAT4 PET in healthy volunteers and patients with lung cancer.
* Determine the acute toxicity of [18F]-C-SNAT4 PET in healthy volunteers and patients with lung cancer.
* Determine whether uptake in [18F]-C-SNAT4 PET imaging is significantly different in tumor and corresponding contralateral noncancer tissue in patients with lung cancer (tested by Wilcoxon test) before the therapy.
* Determine/verify the safety profile of the [18F]-C-SNAT4 radiotracer, as an imaging agent in patients with lung cancer.
* Determine the time of maximal [18F]-C-SNAT4 radiotracer uptake post injection.

ELIGIBILITY:
Inclusion Criteria:

* ANC ≥ 1.5 x 109/L without myeloid growth factor support for 7 days preceding lab assessment
* Hgb ≥ 9 g/dL (90 g/L); < 9 g/dL (< 90 g/L) is acceptable if Hgb corrected to ≥ 9 g/dL (90 g/L) as by growth factor or transfusion prior to PET scan
* Platelet count ≥ 100 x 109/L w/o blood transfusions for 7 days preceding lab assessment
* Bilirubin ≤ 1.5 x upper limit of normal (ULN) except for pts with documented history of Gilbert's disease
* ALT ≤ 2.5 x ULN
* AST ≤ 2.5 x ULN
* Alkaline phosphatase (AP) ≤ 3 x ULN
* If a women of childbearing potential (WCBP): negative early pregnancy test (EPT)
* Karnofsky Performance Status (KPS) ≥ 60
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Has already begun non-surgical therapy for any recurrence, prior to the first [18F]-C-SNAT4 PET/CT scan
* Severe/uncontrolled inter-current illness within the previous 28 days prior to PET scan.
* Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation.
* History of allergic reactions to IV contrasts or reactions attributed to compounds of similar chemical or biological composition to [18F]-C-SNAT4 used in study.
* Pregnant or nursing
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT bore (diameter 70 cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of [18F]-C-SNAT4 | 1 day
  Whole-body [18F]-C-SNAT4 PET scans will be performed at 60 min post intravenous injection of the PET tracer in Group 1 of 5 healthy volunteers

SECONDARY OUTCOMES:
Dosimetry of [18F]-C-SNAT4 | 1 day
  Radiation dosimetry of the [18F]-C-SNAT4 radiotracer will be measured through careful monitoring of each participant's vital signs in Group 1 and group 2. Time-Activity curves will be graphed by measuring activity in various organs using multiple PET/CT scans (1 hour dynamic scan, 1 hour and 2 hours) after tracer injection. Absorbed radiation will be calculated.
Toxicity of [18F]-C-SNAT4 | 7 days
  The acute [18F]-C-SNAT4 toxicity will be assessed as related adverse events, including laboratory abnormalities, that occur within 7 days of the infusion of [18F]-C-SNAT4.
18F]-C-SNAT4 Uptake | 1 day
  The tumor uptake of [18F]-C-SNAT4 PET will be compared with the corresponding contralateral non-cancer tissue in patients with lung cancer before the therapy in Group 2 and 3. SUVmax measurements will be taken from the pre-treatment scan.
The Maximal [18F]-C-SNAT4 Uptake as PET Radiotracer | 1 day
  The time of maximal [18F]-C-SNAT4 radiotracer uptake post-injection will be assessed in Group 2 and 3. Time-Activity Curves (TAC) will be graphed by measuring activity in tumor after tracer injection. The maximal of [18F]-C-SNAT4 radiotracer uptake post-injection in lung cancer patients will be determined from these time activity curves.
[18F]-C-SNAT4 PET Imaging Signal in Responders and Non-responders | 7 days
  The [18F]-C-SNAT4 PET scan signal from pre-therapy to one week after initiation of therapy in Group 3 will be compared both in treatment responders vs. non-responders. SUVmax will be measured in both the pre-treatment and one-week post-initiation of treatment scans.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei H Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No